CLINICAL TRIAL: NCT03222128
Title: Edwards SAPIEN 3 Transcatheter Heart Valve Therapy for Intermediate Risk Patients
Brief Title: PARTNER II Trial: Placement of AoRTic TraNscathetER Valves II - S3 Intermediate
Acronym: PII S3i
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12 PIIS3i
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2018-08-14 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: SAPIEN 3; Transfemoral; Transapical; Transaortic; NovaFlex; TAVI; Aortic Stenosis; THV; Aortic Valve; Transcatheter Heart Valve; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PIIS3i - SAPIEN 3 (Experimental): PIIS3i - SAPIEN 3 is Operable Group
  Interventions: Device: TAVR

INTERVENTIONS:
Device: TAVR — Implantation of the SAPIEN 3

SUMMARY:
The purpose of this trial is to determine the safety and effectiveness of the Edwards SAPIEN 3 transcatheter heart valve and delivery systems which are intended for use in patients with symptomatic, calcific, and severe aortic stenosis, and those with intermediate risk.

DETAILED DESCRIPTION:
This study design consists of PIIS3i cohort.

The PIIS3i cohort is a single arm non-randomized, historical-controlled study. Patients recruited to the treatment arm will receive an Edwards SAPIEN 3 THV with either transfemoral, transapical or transaortic delivery access.

To ensure that patients are of "intermediate" risk, an STS score of 4 - 8% has been selected.

ELIGIBILITY:
Inclusion Criteria

1. Patient has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s and an initial aortic valve area (AVA) of <0.8 cm2 or indexed EOA < 0.5 cm2/m2 Qualifying echo must be within 60 days of the date of the procedure.
2. Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
3. The heart team agrees (and verified in the case review process) that valve implantation will likely benefit the patient.
4. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
5. The study patient agrees to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which will be conducted as a phone follow-up.

Exclusion Criteria:

1. Heart team assessment of inoperability (including examining cardiac surgeon).
2. Complex coronary artery disease

   1. Unprotected left main coronary artery
   2. Syntax score > 32 (in the absence of prior revascularization)
3. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation, or mechanical heart assistance within 30 days of screening evaluation.
4. Need for emergency surgery for any reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1074 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University; Craig Smith, MD, Principal Investigator — Columbia University
Locations (51):
- United States (51):
  - Scripps Green Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Northshore, Evanston, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Indiana University Health-Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc./St. Vincent Heart Center of Indiana, LLC, Indianapolis, Indiana
  - The University of Iowa, Iowa City, Iowa
  - The Jewish Hospital Medical Center, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic-Saint Marys Hospital, Rochester, Minnesota
  - St. Luke's Hospital - Mid America Heart Institute, Kansas City, Missouri
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Northshore Long Island Jewish Health System, New Hyde Park, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - East Carolina Heart Institute at East Carolina University, Greenville, North Carolina
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute at Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Heart, PLLC, Austin, Texas
  - The Heart Hospital Baylor Plano, Dallas, Texas
  - Medical City Dallas, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio (UTHSCSA), San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madhavan MV, Kodali SK, Thourani VH, Makkar R, Mack MJ, Kapadia S, Webb JG, Cohen DJ, Herrmann HC, Williams M, Greason K, Pibarot P, Hahn RT, Jaber W, Xu K, Alu M, Smith CR, Leon MB. Outcomes of SAPIEN 3 Transcatheter Aortic Valve Replacement Compared With Surgical Valve Replacement in Intermediate-Risk Patients. J Am Coll Cardiol. 2023 Jul 11;82(2):109-123. doi: 10.1016/j.jacc.2023.04.049. PMID 37407110
- [Derived] Vincent F, Thourani VH, Ternacle J, Redfors B, Cohen DJ, Hahn RT, Li D, Crowley A, Webb JG, Mack MJ, Kapadia S, Russo M, Smith CR, Alu MC, Leon MB, Pibarot P. Time-of-Day and Clinical Outcomes After Surgical or Transcatheter Aortic Valve Replacement: Insights From the PARTNER Trials. Circ Cardiovasc Qual Outcomes. 2022 Jan;15(1):e007948. doi: 10.1161/CIRCOUTCOMES.121.007948. Epub 2022 Jan 18. PMID 35041482
- [Derived] Herrmann HC, Cohen DJ, Hahn RT, Babaliaros VC, Yu X, Makkar R, McCabe J, Szerlip M, Kapadia S, Russo M, Malaisrie SC, Webb JG, Szeto WY, Kodali S, Thourani VH, Mack MJ, Leon MB. Utilization, Costs, and Outcomes of Conscious Sedation Versus General Anesthesia for Transcatheter Aortic Valve Replacement. Circ Cardiovasc Interv. 2021 Jul;14(7):e010310. doi: 10.1161/CIRCINTERVENTIONS.120.010310. Epub 2021 Jun 16. PMID 34130476
- [Derived] Brener MI, George I, Kosmidou I, Nazif T, Zhang Z, Dizon JM, Garan H, Malaisrie SC, Makkar R, Mack M, Szeto WY, Fearon WF, Thourani VH, Leon MB, Kodali S, Biviano AB. Atrial Fibrillation Is Associated With Mortality in Intermediate Surgical Risk Patients With Severe Aortic Stenosis: Analyses From the PARTNER 2A and PARTNER S3i Trials. J Am Heart Assoc. 2021 Apr 6;10(7):e019584. doi: 10.1161/JAHA.120.019584. Epub 2021 Mar 23. PMID 33754803
- [Derived] Ong G, Pibarot P, Redfors B, Weissman NJ, Jaber WA, Makkar RR, Lerakis S, Gopal D, Khalique O, Kodali SK, Thourani VH, Anwaruddin S, McAndrew T, Zhang Y, Alu MC, Douglas PS, Hahn RT. Diastolic Function and Clinical Outcomes After Transcatheter Aortic Valve Replacement: PARTNER 2 SAPIEN 3 Registry. J Am Coll Cardiol. 2020 Dec 22;76(25):2940-2951. doi: 10.1016/j.jacc.2020.10.032. PMID 33334422
- [Derived] Pibarot P, Ternacle J, Jaber WA, Salaun E, Dahou A, Asch FM, Weissman NJ, Rodriguez L, Xu K, Annabi MS, Guzzetti E, Beaudoin J, Bernier M, Leipsic J, Blanke P, Clavel MA, Rogers E, Alu MC, Douglas PS, Makkar R, Miller DC, Kapadia SR, Mack MJ, Webb JG, Kodali SK, Smith CR, Herrmann HC, Thourani VH, Leon MB, Hahn RT; PARTNER 2 Investigators. Structural Deterioration of Transcatheter Versus Surgical Aortic Valve Bioprostheses in the PARTNER-2 Trial. J Am Coll Cardiol. 2020 Oct 20;76(16):1830-1843. doi: 10.1016/j.jacc.2020.08.049. PMID 33059828
- [Derived] Chen S, Redfors B, O'Neill BP, Clavel MA, Pibarot P, Elmariah S, Nazif T, Crowley A, Ben-Yehuda O, Finn MT, Alu MC, Vahl TP, Kodali S, Leon MB, Lindman BR. Low and elevated B-type natriuretic peptide levels are associated with increased mortality in patients with preserved ejection fraction undergoing transcatheter aortic valve replacement: an analysis of the PARTNER II trial and registry. Eur Heart J. 2020 Feb 21;41(8):958-969. doi: 10.1093/eurheartj/ehz892. PMID 31883339
- [Derived] Summers MR, Leon MB, Smith CR, Kodali SK, Thourani VH, Herrmann HC, Makkar RR, Pibarot P, Webb JG, Leipsic J, Alu MC, Crowley A, Hahn RT, Kapadia SR, Tuzcu EM, Svensson L, Cremer PC, Jaber WA. Prosthetic Valve Endocarditis After TAVR and SAVR: Insights From the PARTNER Trials. Circulation. 2019 Dec 10;140(24):1984-1994. doi: 10.1161/CIRCULATIONAHA.119.041399. Epub 2019 Nov 6. PMID 31690104
- [Derived] Furer A, Chen S, Redfors B, Elmariah S, Pibarot P, Herrmann HC, Hahn RT, Kodali S, Thourani VH, Douglas PS, Alu MC, Fearon WF, Passeri J, Malaisrie SC, Crowley A, McAndrew T, Genereux P, Ben-Yehuda O, Leon MB, Burkhoff D. Effect of Baseline Left Ventricular Ejection Fraction on 2-Year Outcomes After Transcatheter Aortic Valve Replacement: Analysis of the PARTNER 2 Trials. Circ Heart Fail. 2019 Aug;12(8):e005809. doi: 10.1161/CIRCHEARTFAILURE.118.005809. Epub 2019 Aug 1. PMID 31525069
- [Derived] Nazif TM, Chen S, George I, Dizon JM, Hahn RT, Crowley A, Alu MC, Babaliaros V, Thourani VH, Herrmann HC, Smalling RW, Brown DL, Mack MJ, Kapadia S, Makkar R, Webb JG, Leon MB, Kodali SK. New-onset left bundle branch block after transcatheter aortic valve replacement is associated with adverse long-term clinical outcomes in intermediate-risk patients: an analysis from the PARTNER II trial. Eur Heart J. 2019 Jul 14;40(27):2218-2227. doi: 10.1093/eurheartj/ehz227. PMID 31505615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 51 sites in the US
Pre-assignment Details: The As-Treated population was 1074 The Valve-Implanted population was 1069
Period: Overall Study
Arm/Group | PIIS3i - SAPIEN 3
Started | 1074
Valve-Implanted | 1069
Completed (One year follow-up) | 968
Not Completed | 106

BASELINE CHARACTERISTICS:
Arm/Group | PIIS3i - SAPIEN 3
Number analyzed (Participants) | 1074
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 412
  Male | 662
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 5.3 (1.29)
NYHA Classification III/IV [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-V, with the lowest as no limitations and highest unable to carry on any physical activity without discomfort.
  Participants | 780

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of All-cause Death, All Stroke and Aortic Insufficiency (AI) ≥ Moderate
Time Frame: 1 year
Population: AI as a factor in this value; only 964/1069 patients had ECHO data.
Measure: Count of Participants; unit: Participants
Arm/Group | PIIS3i - SAPIEN 3
Number analyzed (Participants) | 964
Participants | 125

2. Secondary Outcome: Composite of All-cause Death, All Stroke, Life Threatening (Disabling)/ Major Bleeding and Major Vascular Complication at 30 Days
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | PIIS3i - SAPIEN 3
Number analyzed (Participants) | 1069
Participants | 196

ADVERSE EVENTS:
Time Frame: The Adverse data collected and reported here are over a period of 1 Year Valve-implant population are noted here.
Description: All Adverse Events are site-reported.
Arm/Group | PIIS3i - SAPIEN 3
All-Cause Mortality (participants affected / at risk) | 75/1069
Serious Adverse Events (participants affected / at risk) | 592/1069
Other Adverse Events (participants affected / at risk) | 861/1069
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIIS3i - SAPIEN 3 (N=1069)
Abnormal lab value (Metabolism and nutrition disorders) | 22 (26)
Access site and access related vascular injury - Dissection (Vascular disorders) | 11 (11)
Access site and access related vascular injury - Distal embolization (noncerebral) from vascular sou (Vascular disorders) | 1 (1)
Access site and access related vascular injury - Failure of percutaneous access site closure (Injury, poisoning and procedural complications) | 8 (8) — resulting in intervention
Access site and access related vascular injury - Hematoma (Vascular disorders) | 5 (5)
Access site and access related vascular injury - Other (Vascular disorders) | 8 (8)
Access site and access related vascular injury - Perforation (Vascular disorders) | 4 (4)
Access site and access related vascular injury - Pseudoaneurysm (Vascular disorders) | 4 (4)
Access site and access related vascular injury - Rupture (Vascular disorders) | 1 (1)
Access site and access related vascular injury - Stenosis (Vascular disorders) | 5 (5)
Access site and access related vascular injury - Ventricular rupture (Apical rupture) (Vascular disorders) | 2 (2)
Anemia/Hemolytic anemia (Blood and lymphatic system disorders) | 25 (29)
Anesthesia related complication - Confusion (Injury, poisoning and procedural complications) | 1 (1)
Anesthesia related complication - Other (Injury, poisoning and procedural complications) | 1 (1)
Angina/Cardiac chest pain (Cardiac disorders) | 16 (17)
Aortic Valve Stenosis (Cardiac disorders) | 2 (2)
Aortic insufficiency/Regurgitation PV leak - Non structural dysfunction (Cardiac disorders) | 7 (7)
Aortic insufficiency/Regurgitation PV leak - Structural dysfunction (General disorders) | 1 (1)
Aortic insufficiency/Regurgitation non valvular cause (General disorders) | 1 (1)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 195 (216)
Bleeding - Hemorrhage (Injury, poisoning and procedural complications) | 111 (134)
Cardiac arrest (Cardiac disorders) | 17 (17)
Cardiac tamponade/Pericardial effusion (Cardiac disorders) | 14 (14)
Cardiogenic shock (Cardiac disorders) | 2 (3)
Carotid artery disease (Nervous system disorders) | 5 (5)
Coronary artery disease/Coronary ischemia (Cardiac disorders) | 8 (11)
Coronary flow obstruction/Transvalvular flow disturbance (Cardiac disorders) | 1 (1)
Delirium (Psychiatric disorders) | 3 (3)
Device migration/malposition requiring intervention (Injury, poisoning and procedural complications) | 3 (3)
Edema (Ear and labyrinth disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (3)
Exercise intolerance or weakness (Metabolism and nutrition disorders) | 2 (2)
Gastro Intestinal event - Non-hemorrhagic (Gastrointestinal disorders) | 31 (33)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 17 (17)
Heart failure/CHF/Low output failure (Cardiac disorders) | 76 (96)
Hemolysis (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (10)
Hypotension (Vascular disorders) | 11 (11)
Infection - Access site infection (Infections and infestations) | 4 (4)
Infection - Bacteremia (Infections and infestations) | 5 (5)
Infection - Endocarditis (Infections and infestations) | 8 (8)
Infection - Other (Infections and infestations) | 26 (27)
Infection - Respiratory infection (Infections and infestations) | 55 (63)
Infection - Sepsis (Infections and infestations) | 28 (29)
Infection - Urinary tract infection (Infections and infestations) | 20 (21)
Ischemia (Investigations) | 8 (10)
Myocardial Infarction (Cardiac disorders) | 13 (15)
Mental state change (not neurological) - Confusion (Investigations) | 5 (5)
Mental state change (not neurological) - Dementia (Investigations) | 2 (2)
Mental state change (not neurological) - Depression (Investigations) | 2 (2)
Miscellaneous - Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17)
Miscellaneous - Drug reaction (Investigations) | 2 (2)
Miscellaneous - Fall (Injury, poisoning and procedural complications) | 23 (25)
Miscellaneous - Other (General disorders) | 15 (15)
Miscellaneous - Suicide (Social circumstances) | 1 (1)
Mitral valve injury or insufficiency (Cardiac disorders) | 3 (3)
Multi organ failure (General disorders) | 1 (1)
Musculoskeletal - Fracture (Injury, poisoning and procedural complications) | 33 (36)
Musculoskeletal - Pain (Musculoskeletal and connective tissue disorders) | 25 (25)
Neurological - Change in level of consciousness (Nervous system disorders) | 1 (1)
Neurological - Cognitive impairment (Nervous system disorders) | 2 (2)
Neurological - Dysphasia/Aphasia (Nervous system disorders) | 1 (1)
Neurological - Hemiparesis (One sided body weakness) (Nervous system disorders) | 1 (1)
Neurological - Hemorrhagic stroke (Nervous system disorders) | 8 (8)
Neurological - Ischemic stroke (Nervous system disorders) | 24 (25)
Neurological - Other (Nervous system disorders) | 6 (7)
Neurological - Other new neurological sign consistent with stroke (Nervous system disorders) | 1 (1)
Neurological - TIA (Nervous system disorders) | 10 (12)
Neurological - Undetermined stroke (Nervous system disorders) | 7 (8)
Pericarditis (Cardiac disorders) | 1 (1)
Renal insufficiency or renal failure (Renal and urinary disorders) | 31 (34)
Respiratory event - Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory event - Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory event - Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Respiratory event - Other (Respiratory, thoracic and mediastinal disorders) | 17 (18)
Respiratory event - Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory event - Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory event - Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Respiratory event - Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 32 (37)
Syncope (Vascular disorders) | 14 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (15)
Thromboembolic event (Vascular disorders) | 13 (13)
Unknown cause of death (General disorders) | 5 (5)
Valve thrombosis (Vascular disorders) | 1 (1)
Vascular complication - Non-access related (Vascular disorders) | 16 (18)
Other (General disorders) | 38 (41)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIIS3i - SAPIEN 3 (N=1069)
Abnormal lab value (Investigations) | 144 (186)
Anemia/Hemolytic anemia (Blood and lymphatic system disorders) | 128 (140)
Aortic insufficiency/Regurgitation PV leak - Non structural dysfunction (Cardiac disorders) | 55 (55)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 299 (357)
Bleeding - Hemorrhage (Vascular disorders) | 212 (240)
Gastro Intestinal event - Non-hemorrhagic (Gastrointestinal disorders) | 66 (77)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 83 (88)
Heart failure/CHF/Low output failure (Cardiac disorders) | 95 (101)
Hypertension (Vascular disorders) | 57 (59)
Hypotension (Vascular disorders) | 63 (68)
Infection - Other (Infections and infestations) | 55 (62)
Infection - Urinary tract infection (Infections and infestations) | 87 (101)
Miscellaneous - Fall (Injury, poisoning and procedural complications) | 70 (81)
Miscellaneous - Other (Investigations) | 65 (72)
Musculoskeletal - Pain (Musculoskeletal and connective tissue disorders) | 81 (94)
Renal insufficiency or renal failure (Renal and urinary disorders) | 117 (134)
Respiratory event - Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 63 (67)
Thrombocytopenia (Blood and lymphatic system disorders) | 101 (101)
Other (Investigations) | 111 (136)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes